CLINICAL TRIAL: NCT01204476
Title: Phase I Study of Anti-IGF-1R Monoclonal Antibody, IMC-A12, and mTOR Inhibitor, Everolimus, in Advanced Low to Intermediate Grade Neuroendocrine Carcinoma
Brief Title: Cixutumumab, Everolimus, and Octreotide Acetate in Treating Patients With Advanced Low to Intermediate Grade Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-02196; NCI-2010-02196 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000685267; 2009-0734; 2009-0734 (Other: M D Anderson Cancer Center); 8354 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Gastrin-Producing Neuroendocrine Tumor; Lung Carcinoid Tumor; Metastatic Digestive System Neuroendocrine Tumor G1; Pancreatic Glucagonoma; Pancreatic Insulinoma; Pancreatic Polypeptide Tumor; Paraganglioma; Recurrent Digestive System Neuroendocrine Tumor G1; Recurrent Merkel Cell Carcinoma; Recurrent Pancreatic Neuroendocrine Carcinoma; Regional Digestive System Neuroendocrine Tumor G1; Somatostatin-Producing Neuroendocrine Tumor; Stage III Merkel Cell Carcinoma; Stage IV Merkel Cell Carcinoma; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Zollinger-Ellison Syndrome; Glucagonoma; Insulinoma; Paraganglioma; Carcinoma, Merkel Cell; Somatostatinoma; Carcinoma, Medullary | interventions — cixutumumab; Everolimus; Octreotide; Acetates; Salts

ARMS (1):
- Treatment (cixutumumab, octreotide acetate, everolimus) (Experimental): Patients receive cixutumumab IV over 60-90 minutes and octreotide acetate IM on day 1 and everolimus PO QD on days 1-21. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Drug: Everolimus; Other: Laboratory Biomarker Analysis; Drug: Octreotide Acetate; Other: Pharmacological Study

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Octreotide Acetate — Given IM
  Other Names: D-Phenylalanyl-L-cysteinyl-L-phenylalanyl-D-tryptophyl-L-lysyl-L-threonyl-N-[(1R,2R)-2-hydroxy-1-(hyroxymethyl)propyl]-L-cysteinamide, Cyclic (2->7)-disulfide, Acetate (Salt); Longastatin; Longastatina; Samilstin; Sandostatin; Sandostatin Lar Depot; Sandostatina; Sandostatine; SMS 201-995; SMS 201-995 AC
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of cixutumumab when given together with everolimus and octreotide acetate in treating patients with advanced low- or intermediate-grade neuroendocrine cancer. Monoclonal antibodies, such as cixutumumab, may find tumor cells and help carry tumor-killing substances to them. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Octreotide acetate may interfere with the growth of tumor cells and slow the growth of neuroendocrine cancer. Giving cixutumumab together with everolimus and octreotide acetate may be a better treatment for neuroendocrine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To recommend a phase 2 dose for the combination of IMC-A12 (cixutumumab) and everolimus, given with octreotide long-acting release (LAR) (octreotide acetate), in patients with advanced neuroendocrine tumors.

II. To describe the pharmacokinetics of IMC-A12 given once every 21 days in combination with everolimus and octreotide LAR.

III. To evaluate pharmacodynamic markers in blood, and tumor tissue.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of IMC-A12 and everolimus with octreotide LAR.

II. To explore the anti-tumor activity of the combination of IMC-A12 and everolimus as defined by Response Evaluation Criteria in Solid Tumors (RECIST) response rate and progression-free survival (PFS).

TERTIARY OBJECTIVES:

I. To explore baseline molecular marker and drug-induced molecular marker changes that may predict clinical outcome.

OUTLINE: This is a dose-escalation study of cixutumumab.

Patients receive cixutumumab intravenously (IV) over 60-90 minutes and octreotide acetate intramuscularly (IM) on day 1 and everolimus orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study
* Patients must have histologically or cytologically confirmed low or intermediate grade neuroendocrine carcinoma, for which standard curative measures do not exist; patients with neuroendocrine tumors associated with multiple endocrine neoplasia type 1 (MEN1) syndrome will be eligible
* Patients must have disease that is amenable to computed tomography (CT) or ultrasound (U/S) guided biopsies; patients must agree to undergo 2 biopsies; the disease identified for biopsy cannot be the only site of measurable disease
* Patients must be registered in the M.D. Anderson Cancer Center (MDACC) institutional database prior to treatment with study drug
* Zubrod performance status of 0 or 1
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Hemoglobin > 9 g/dL; eligibility level for hemoglobin may be reached by transfusion
* Platelets > 100,000/mcL
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 1.5 X institutional ULN (5 x ULN if liver function tests [LFT] elevations due to liver metastases)
* Creatinine =< 1.5 X institutional ULN OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The patient must have fasting serum glucose =< 1.2 X upper limit of normal
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN; NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Women of child-bearing potential and men must agree to use adequate contraception from the time of study enrollment continuing for the duration of study therapy and for 3 months after the last dose of IMC-A12 and/or everolimus; oral, implantable, or injectable contraceptives are not considered effective for this study; if barrier contraceptives are being used, these must be continued for the specified time by both sexes; women are considered to be of child-bearing potential if they have not undergone surgical sterilization (laparoscopic tubal ligation, hysterectomy, bilateral salping-oophorectomy) or have not reached menopause, defined as amenorrhea persisting for at least twelve consecutive months; men of any age are considered to be fertile unless they have undergone bilateral vasectomy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; if the subject becomes pregnant while on study, she must discontinue study treatment
* Negative pregnancy test (serum beta-human chorionic gonadotropin [HCG]) within 7 days of starting study treatment is required in women of childbearing potential; neuroendocrine tumor (NET) patients with positive beta-HCG are eligible if pregnancy can be excluded by lack of expected doubling of beta-HCG; the usual beta-HCG doubling time is every 2 days during the first 4 weeks of pregnancy and lengthens to every 3 ½ days by weeks 6 to 7; patients can also be eligible if pregnancy can be excluded by vaginal ultrasound in consultation with Obstetrics/Gynecology
* Patients must have at least one measurable site of disease according to RECIST that has not been previously irradiated; if the patient has had previous radiation to the target lesion(s), there must be evidence of progression in the lesion(s) since the radiation
* Prior radiation therapy is permitted; a recovery period of at least 4 weeks after completion of radiotherapy is required prior to enrollment
* Patients may have received prior systemic anti-neoplastic therapy (except prior mammalian target of rapamycin [mTOR] inhibitors or agents targeting insulin-like growth factor 1 receptor [IGF1R]); there are no limitations on the number of prior regimens; at least 28 days must have elapsed since last treatment
* Patients not on anticoagulation must have international normalized ratio (INR) =< 1.5; patients on full-dose anticoagulation (warfarin or low molecular weight heparin) are eligible provided that both of the following criteria are met:

  * The patient has an in-range INR (between 2 and 3) on a stable (no change in the 2 weeks prior to registration) dose of oral anticoagulant or on a stable (no change in the prior 2 weeks) dose of low molecular weight heparin
  * The patient has no active bleeding or known pathological condition that carries a high risk of bleeding such as varices

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring parenteral therapy at the time of study registration
  * Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C); note: a detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients
  * Symptomatic congestive heart failure resulting in a resting oxygen saturation of < 92% on room air
  * Unstable angina or pectoris myocardial infarction within 6 months of start of study drug
  * Serious uncontrolled cardiac arrhythmia
  * Known severely impaired lung function as defined as spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or oxygen saturation that is 88% or less at rest on room air; pulmonary function test (PFT) is not required at study entry
* A known history of human immunodeficiency virus (HIV) seropositivity
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; pregnant women are excluded from the study; breastfeeding women should be excluded
* Patients with a known history of allergic reactions and/or hypersensitivity attributed compounds of similar chemical or biologic composition to IMC-A12, everolimus or other rapamycins (sirolimus, temsirolimus)
* Known history of brain or leptomeningeal metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Patients who have had hormonal therapy (other than replacement) within 4 weeks prior to entering the study
* Not recovered from adverse events related to previous treatment (excluding alopecia) to active Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1
* With the exception of tumor common to a single genetic cancer syndrome (i.e. MEN1, multiple endocrine neoplasia type 2 [MEN2], von Hippel-Lindau [vHL], tuberous sclerosis complex [TSC] etc), patients with evidence of more than one active malignancy are excluded; active malignancy is defined as the presence of primary, regional nodal, or distant metastatic neoplasm that has not undergone definitive therapy
* The patient has poorly controlled diabetes mellitus; patients with a history of diabetes mellitus are allowed to participate, providing that their blood glucose is within 1.2 X institutional upper limit of normal and that they are on a stable dietary or therapeutic regimen for this condition
* Patients who have received prior treatment with IMC-A12, everolimus, other agents targeting the insulin-like growth factor receptor (IGFR) or an mTOR inhibitor (sirolimus, temsirolimus, everolimus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) for the combination of cixutumumab and everolimus with octreotide acetate | 21 days
  Analysis will be performed using a patient summary of the number of cycles of study drug administered by initial dose level, and will be presented including a flag for DLTs which occurred during course 1. The recommended Phase II dose will also be presented.
Pharmacodynamic markers in blood and tumor tissue | Up to day 1 of course 4
  Descriptive statistics for the changes from baseline in blood and tissue biomarkers will be presented by response category in an attempt to characterize these changes with respect to efficacy.
Pharmacokinetic parameters | Pre-dose and day 1 of courses 1-7
  Descriptive statistics will be used for plasma drug concentration data. Calculated parameters will include maximum concentration and minimum concentration.
Safety profile of cixutumumab and everolimus with octreotide acetate among patients with advanced neuroendocrine tumors, defined by the incidence of adverse events | Up to 30 days after completion of study treatment
  Safety data will be tabulated for all patients who receive any amount of study medication. These data will include adverse events and laboratory parameters. Adverse events will be tabulated by body system, preferred term, severity and relation to treatment. The tabulation of adverse events will be done using the CTCAE version 4.0.

SECONDARY OUTCOMES:
Anti-tumor activity as determined by RECIST | Up to 30 days after completion of study treatment

OTHER OUTCOMES:
Changes in drug-induced molecular markers | Baseline to up to day 1 of course 4
Changes in molecular markers | Baseline to up to day 1 of course 4

CONTACTS AND LOCATIONS:
Overall Officials: James Yao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Dasari A, Phan A, Gupta S, Rashid A, Yeung SC, Hess K, Chen H, Tarco E, Chen H, Wei C, Anh-Do K, Halperin D, Meric-Bernstam F, Yao J. Phase I study of the anti-IGF1R antibody cixutumumab with everolimus and octreotide in advanced well-differentiated neuroendocrine tumors. Endocr Relat Cancer. 2015 Jun;22(3):431-41. doi: 10.1530/ERC-15-0002. Epub 2015 Apr 21. PMID 25900182